CLINICAL TRIAL: NCT00122720
Title: The Effect of Darbepoetin Alfa Treatment Upon the Rehabilitation Following Planned Surgery for Colorectal Cancer
Brief Title: The Effect of Darbepoetin Upon Rehabilitation for Colorectal Cancer Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Herning Hospital (Other)
Collaborators: Amgen (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 2612-2277
Record Dates: First submitted 2005-07-20; First posted 2005-07-22 (Estimated); Last update posted 2006-07-07 (Estimated); Status verified 2006-01

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; erythropoietin; rehabilitation; physical capacity
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Darbepoetin alfa

INTERVENTIONS:
Drug: Darbepoetin Alfa

SUMMARY:
The study is investigating whether randomization to perioperative darbepoetin alfa treatment improves the rehabilitation following surgery for colonic and rectal cancer.

DETAILED DESCRIPTION:
Major surgery elicits a metabolic stress response that is followed by a loss of body mass, fatigue, and an impaired physical performance including a reduced work capacity.

To perform ordinary daily activities many elderly people exert close to their maximum physical capacity, and even a small reduction of performance capacity may cause significant impairment in physical and social activity. Postoperative decline in strength and work capacity may thus cause previously independent living persons to become dependent upon assistance from others. Hence, it is important to avoid the postoperative reduction of physical performance and to minimize postoperative fatigue.

It has been shown that Erythropoietin treatment reduces the need for blood transfusions in patients undergoing planned colonic surgery. However, the effect of Erythropoietin treatment upon postoperative rehabilitation has not yet been studied.

Therefore the main hypothesis in this study is that perioperative treatment with Darbepoetin Alfa would improve the physical capacity in aspects by reducing postoperative fatigue and improve work capacity, balance and quality of life compared to placebo treatment. Furthermore, the researchers expect Darbepoetin treated patients to have fewer perioperative complications and less need for blood transfusions.

ELIGIBILITY:
Inclusion Criteria:

* Planned colonic and rectal surgery because of presumed cancer disease in the colon and rectum

Exclusion Criteria:

* Psychiatric disease or dementia
* Diseases, that renders participation in the study impossible
* Thromboembolic disease within the last three months
* Dysregulated hypertension (systolic blood pressure>175 mmHg and/or diastolic blood pressure>105 mmHg)
* Other diseases or causes that will contraindicate treatment with Darbepoetin Alfa
* Other diseases or causes that will contraindicate further treatment with Darbepoetin Alfa
* Patients that preoperatively and/or four days postoperatively have a hemoglobin concentration > 14 g/dl
* Former cancer disease
* Disseminated cancer disease
* Rectal cancer stage T4

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2003-06; Study Completion 2006-01

PRIMARY OUTCOMES:
The functional capacity measured by postoperative fatigue, work capacity, balance, and quality of life

SECONDARY OUTCOMES:
Muscular strength
Weight
Body composition
Blood transfusion
Postoperative complications

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte B Norager, M.D., Principal Investigator — Surgical Research Department, Herning Hospital, Gl. Landevej 61, DK-7400 Herning
Locations (5):
- Denmark (5):
  - Surgical Department, Aarhus University Hospital, Aarhus, Aarhus
  - Surgical Department, Middelfart Hospital, Middelfart, Fyn
  - Surgical Department, Odense University Hospital, Odense, Fyn
  - Surgical Department, Svendborg Hospital, Svendborg, Fyn
  - Surgical Department, Herning Hospital, Herning, Ringkobing